CLINICAL TRIAL: NCT07250633
Title: A Phase 1, Open-Label, Non-randomized, Single Dose, Safety, Tolerability, and Pharmacokinetic Study of Vorasidenib Administered to Participants With Severe Hepatic Impairment and Matched-Participants With Normal Hepatic Function
Brief Title: Pharmacokinetic Study of Vorasidenib in Severe Hepatically Impaired and Matched-Control Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (I.R.I.S.) (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: S95032-223
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Severe Hepatic Impairment; Normal Hepatic Function
MeSH Terms: interventions — vorasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants with Severe Hepatic Impairment (HI) (Experimental)
  Interventions: Drug: Vorasidenib 20mg
- Matched-Participants with Normal Hepatic Function (Experimental)
  Interventions: Drug: Vorasidenib 20mg

INTERVENTIONS:
Drug: Vorasidenib 20mg — Vorasidenib 20mg will be taken by mouth on Day 1

SUMMARY:
The objective of this study is to evaluate the pharmacokinetics, safety, and tolerability of one dose of vorasidenib in participants with severe impaired hepatic function compared to participants with normal hepatic function. The study includes a screening phase, a treatment period, and a follow-up period. During the first part of the treatment period, from Day 1 through Day 4, participants will remain in-house in the clinical research unit. In the second part of the treatment period, from Day 5 through Day 43, participants can go home but may also choose to remain in-house. The entire study, including screening and follow-up, will last up to 77 days. Participants may undergo blood tests, heart tests (electrocardiogram (ECG)), vital sign checks, and physical exams.

ELIGIBILITY:
Inclusion Criteria:

Participants with hepatic impairment:

* Diagnosis of cirrhosis due to parenchymal liver disease
* Considered to have a Child-Pugh score of 10 to 15, consistent with severe HI, and a documented medical history of liver disease. Participants must be clinically stable (no acute episodes of illness due to deterioration in hepatic function) for at least 1 month prior to screening and are likely to remain stable throughout the study.
* Grade 0 or Grade 1 hepatic encephalopathy considered stable per Investigator assessment without exacerbation within the 6 months prior to screening.
* Currently on a stable medication regimen, defined as not starting new drug(s) or significantly changing drug dosage(s) within 14 days preceding Day 1.
* Non-hepatic abnormal laboratory values must be not clinically significant as judged by the Investigator (or designee) and the study medical monitor.
* Anemia secondary to hepatic disease is acceptable if hemoglobin is ≥ 9 g/dL and anemia symptoms are not clinically significant. Platelet count must be ≥ 35,000 platelets.
* QT interval corrected for heart rate using Fridericia's formula (QTcF) of ≤ 480 msec.

Matched-control participants:

* Healthy, with normal hepatic function with a Child-Pugh score below 5.
* Resting blood pressure of 90 to 140 mmHg (systolic) and 40 to 90 mmHg (diastolic).
* QTcF of ≤ 450 msec.
* Participant must match hepatically impaired participants with respect to sex, race, age (±10 years), smoking status (smoke or vape ≤ 10 cigarettes/day), and body mass index (±20%).

Exclusion Criteria for all participants:

* Women of childbearing potential (WOCBP) who are pregnant, lactating, or planning to become pregnant within 90 days after the dose of vorasidenib.
* The participant is using hormonal contraceptives
* Use of any other investigational drug or device within 30 days (or 5 half-lives if known, whichever is longer) before the dose of vorasidenib
* Consumption of any nutrients known to modulate CYP450 enzymes activity (e.g., grapefruit or grapefruit juice, pomelo juice, star fruit, Seville [blood] orange products) within 14 days before vorasidenib administration.
* Consumption of alcohol-containing foods or beverages or caffeine- or xanthine-containing foods or beverages (including, but not limited to, teas [including decaffeinated teas], coffees [including decaffeinated coffees], colas [including decaffeinated colas], energy drinks, gum containing caffeine, and chocolate (including foods and beverages containing chocolate) within 48 hours prior to admission
* Any history (within 5 years prior to screening) or presence of malignancy, except for adequately treated basal cell and squamous cell carcinoma of the skin
* History within the previous 12 months of alcohol consumption exceeding 2 standard drinks per day on average (1 standard drink = 12 oz beer, 5 oz wine, or 1.5 oz spirits)
* In the opinion of the Investigator, the participant is not suitable for entry into the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Through the end of the treatment period (approximately 43 days)
Area under the plasma concentration-time curve (AUC) from time 0 to the last quantifiable concentration (AUC0-t) | Through the end of the treatment period (approximately 43 days)
AUC from time 0 extrapolated to infinity (AUC0-inf) | Through the end of the treatment period (approximately 43 days)
Time to reach Cmax (Tmax) | Through the end of the treatment period (approximately 43 days)
Apparent terminal elimination half-life (t1/2) | Through the end of the treatment period (approximately 43 days)
Apparent oral clearance (CL/F) | Through the end of the treatment period (approximately 43 days)
Apparent volume of distribution (Vz/F) | Through the end of the treatment period (approximately 43 days)
Apparent terminal elimination rate constant (Kel) | Through the end of the treatment period (approximately 43 days)

SECONDARY OUTCOMES:
Number of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Through the end of the study (approximately 50 days)
Number of participants experiencing clinically significant changes in laboratory assessments, vital signs, ECG results, or physical examination findings | Through the end of the study (approximately 50 days)

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorization in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.